CLINICAL TRIAL: NCT03786783
Title: A Pilot Induction Regimen Incorporating Chimeric 14.18 Antibody (ch14.18, Dinutuximab) (NSC# 764038) and Sargramostim (GM-CSF) for the Treatment of Newly Diagnosed High-Risk Neuroblastoma
Brief Title: Dinutuximab, Sargramostim, and Combination Chemotherapy in Treating Patients With Newly Diagnosed High-Risk Neuroblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-03732; NCI-2018-03732 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANBL17P1 (Other: Children's Oncology Group); ANBL17P1 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2018-12-24; First posted 2018-12-26 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Ganglioneuroblastoma; High Risk Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma | interventions — Stem Cell Transplantation; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Dexrazoxane; Razoxane; dinutuximab; Doxorubicin; Etoposide; Congresses as Topic; Radiation; Isotretinoin; Melphalan; sargramostim; Colony-Stimulating Factors; Thiotepa; Topotecan; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment(chemotherapy, dinutuximab, sargramostim, ASCT, EBRT) (Experimental): See Detailed Description
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Dexrazoxane; Biological: Dinutuximab; Drug: Doxorubicin; Drug: Etoposide; Radiation: External Beam Radiation Therapy; Drug: Isotretinoin; Drug: Melphalan; Biological: Sargramostim; Drug: Thiotepa; Drug: Topotecan; Drug: Vincristine

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Dexrazoxane — Given IV
  Other Names: 2, 6-Piperazinedione, 4,4'-propylenedi-, (P)- (8CI); 2,6-Piperazinedione, 4, 4'-(1-methyl-1,2-ethanediyl)bis-, (S)- (9CI); ADR 529; ADR-529; ADR529; ICRF 187; ICRF-187; ICRF187; Razoxane (+)-form; Soluble ICRF (L-isomer)
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Topotecan — Given IV
  Other Names: Hycamptamine; Topotecan Lactone
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II pilot trial studies the side effects and how well dinutuximab and sargramostim work when combined with chemotherapy in patients with high-risk neuroblastoma. Immunotherapy with monoclonal antibodies, such as dinutuximab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread. Sargramostim helps the body produce normal infection-fighting white blood cells. These cells also help the dinutuximab work better. Giving chemotherapy before a stem cell transplant, with drugs such as cisplatin, etoposide, vincristine, doxorubicin, cyclophosphamide, thiotepa, melphalan, etoposide, carboplatin, topotecan, and isotretinoin, helps kill cancer cells that are in the body and helps make room in a patient's bone marrow for new blood-forming cells (stem cells). Giving dinutuximab and sargramostim with combination chemotherapy may work better than combination chemotherapy alone in treating patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and tolerability of administering ch14.18 (dinutuximab) and sargramostim (GM-CSF) in combination with a multi-agent chemotherapy regimen during cycles 3-5 of the Induction phase for patients with newly-diagnosed high-risk neuroblastoma.

SECONDARY OBJECTIVE:

I. To describe the response rates, event-free survival (EFS) and overall survival (OS) for patients receiving the combination of standard Induction chemotherapy and ch14.18 (dinutuximab) followed by tandem transplant, radiation therapy, and post-consolidation immunotherapy.

EXPLORATORY OBJECTIVES:

I. To describe the clinical relevance of naturally occurring anti-glycan antibodies in patients receiving ch14.18 (dinutuximab).

II. To describe the clinical relevance of natural killer (NK) receptor NKp30 isoforms in patients receiving ch14.18 (dinutuximab).

III. To describe the association between host factors, including human anti-chimeric antibodies (HACA), and response to protocol therapy.

IV. To describe the immune environment (gene expression; immune effector cells, activities and signaling molecules; immune target expression) during and following treatment.

V. To describe the association between levels of circulating GD2, and tumor cell GD2 expression with response to therapy.

OUTLINE:

INDUCTION CYCLES 1-2 (21 days): Patients receive cyclophosphamide intravenously (IV) over 15-30 minutes and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.

INDUCTION CYCLE 3: Patients receive cisplatin IV over 1 hour on days 1-3, etoposide IV over 2 hours on days 1-3, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim subcutaneously (SC) on day 6 or 7 of a 21-day cycle.

INDUCTION CYCLE 4: Patients receive vincristine IV over 1 minute on day 1, doxorubicin IV over 1-15 minutes on days 1-2, cyclophosphamide IV over 1 hour on days 1-2, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim SC on day 6 or 7 of a 21-day cycle.

INDUCTION CYCLE 5: Patients receive cisplatin IV over 1 hour on days 1-3, etoposide IV over 2 hours on days 1-3, dinutuximab IV over 10-20 hours on days 2-5, and sargramostim SC on day 6 or 7 of a 21-day cycle.

Patients may undergo surgery after the fourth or fifth cycle of Induction at the discretion of treating doctor. Patients with stable disease or better tumor response at the end of Induction proceed to Consolidation. Consolidation treatment begins between 4 and 6 weeks from the start date of Induction chemotherapy cycle 5. For patients who have surgical resection delayed until after Induction chemotherapy cycle 5, Consolidation starts within 4 weeks from the date of surgery.

CONSOLIDATION #1: Patients receive thiotepa IV over 2 hours on days -7 to -5 and cyclophosphamide IV over 1 hour on days -5 to -2. Patients then undergo autologous stem cell transplant (ASCT) on day 0.

CONSOLIDATION #2: Patients receive melphalan IV over 30 minutes on days -7 to -5, etoposide IV over 24 hours on days -7 to -4, and carboplatin IV over 24 hours on days -7 to -4. Patients then undergo ASCT on day 0.

RADIATION THERAPY: Beginning 42-80 days following Consolidation #2, patients receive external beam radiation therapy (EBRT) daily for up to 20 days.

Patients then receive post-Consolidation therapy starting at least 1 week following radiation therapy.

POST-CONSOLIDATION CYCLES 1-5: Patients receive sargramostim SC on days 1-14, dinutuximab IV over 10-20 hours on days 4-7, and isotretinoin orally (PO) twice daily (BID) on days 11-24. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

POST-CONSOLIDATION CYCLE 6: Patients receive isotretinoin PO BID on days 15-28 of a 28-day cycle.

After completion of study treatment, patients are followed up at months 3, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, and 60.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on ANBL00B1 or APEC14B1 prior to enrollment on ANBL17P1.
* Patients must have a diagnosis of neuroblastoma or ganglioneuroblastoma (nodular) verified by tumor pathology analysis or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites. The following disease groups are eligible:

  * Patients with International Neuroblastoma Risk Group (INRG) stage M disease are eligible if found to have either of the following features:

    * MYCN amplification (> 4-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features; OR
    * Age > 547 days regardless of biologic features;
  * Patients with INRG stage MS disease with MYCN amplification
  * Patients with INRG stage L2 disease with MYCN amplification
  * Patients > 547 days of age initially diagnosed with INRG stage L1, L2 or MS disease who progress to stage M without prior chemotherapy may enroll within 4 weeks of progression to stage M.
  * Patients >= 365 days of age initially diagnosed with MYCN amplified INRG stage L1 disease who progress to stage M without systemic therapy may enroll within 4 weeks of progression to stage M.
* Patients initially recognized to have high-risk disease must have had no prior systemic therapy (other than topotecan/cyclophosphamide initiated on an emergent basis and within allowed timing as described).
* Patients observed or treated with a single cycle of chemotherapy per a low or intermediate risk neuroblastoma regimen (e.g., as per ANBL0531, ANBL1232 or similar) for what initially appeared to be non-high risk disease but subsequently found to meet the criteria will also be eligible.
* Patients who receive localized emergency radiation to sites of life-threatening or function-threatening disease prior to or immediately after establishment of the definitive diagnosis will be eligible.
* Creatinine clearance (CrCl) or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/sex as follows:

  * Age 1 month to < 6 months (male 0.4 mg/dL, female 0.4 mg/dL)
  * Age 6 months to < 1 year (male 0.5 mg/dL, female 0.5 mg/dL)
  * Age 1 to < 2 years (male 0.6 mg/dL, female 0.6 mg/dL)
  * Age 2 to < 6 years (male 0.8 mg/dL, female 0.8 mg/dL)
  * Age 6 to < 10 years (male 1 mg/dL, female 1 mg/dL)
  * Age 10 to < 13 years (male 1.2 mg/dL, female 1.2 mg/dL)
  * Age 13 to < 16 years (male 1.5 mg/dL, female 1.4 mg/dL)
  * Age >= 16 years (male 1.7 mg/dL, female 1.4 mg/dL) (within 7 days prior to enrollment).
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment).
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 10 x ULN. For the purposes of this study, ULN for ALT is 45 IU/L (within 7 days prior to enrollment).
* Shortening fraction of >= 27% by echocardiogram (within 7 days prior to enrollment).
* Ejection fraction of >= 50% by echocardiogram or radionuclide angiogram (within 7 days prior to enrollment).
* No known contraindication to peripheral blood stem cell (PBSC) collection. Examples of contraindications might be a weight or size less than the collecting institution finds feasible, or a physical condition that would limit the ability of the child to undergo apheresis catheter placement (if necessary) and/or the apheresis procedure.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patients >18 months of age with INRG stage L2, MYCN non-amplified, regardless of additional biologic features.
* Patients with bone marrow failure syndromes.
* Patients that are >= 12 and =< 18 months of age with INRG stage M and all 3 favorable biologic features (i.e., non-amplified MYCN, favorable pathology, and deoxyribonucleic acid [DNA] index > 1) are not eligible.
* Patients on immunosuppressive medications (e.g. tacrolimus, cyclosporine, corticosteroids for reasons other than prevention/treatment of allergic reactions, adrenal replacement therapy, etc.) are not eligible.
* Female patients who are pregnant are ineligible since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
* Lactating females who plan to breastfeed their infants.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method during study therapy and for two months after the last dose of ch14.18 (dinutuximab) are not eligible.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-09-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Federico, Principal Investigator — Children's Oncology Group
Locations (10):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
- Starship Children's Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with newly diagnosed high-risk Neuroblastoma enrolled between 1/14/2019 and 9/4/2020 across 10 institutions.
Groups:
- Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT): Patients receive 5 cycles of Induction chemotherapy including cyclophosphamide, topotecan, cisplatin, etoposide, dinutuximab, sargramostim, vincristine, and doxorubicin. Patients may undergo surgery after Cycle 4 or 5 of Induction at the discretion of treating doctor. Patients with stable disease or better tumor response at end of Induction proceed to Consolidation. Consolidation treatment begins between 4-6 weeks from the start date of Induction cycle 5. For patients who have surgical resection delayed until after Induction cycle 5, Consolidation starts within 4 weeks from the date of surgery. Patients then undergo 2 cycles of Consolidation including thiotepa, cyclophosphamide, melphalan, etoposide, and carboplatin, followed by Radiation therapy beginning 42-80 days following Consolidation Cycle #2. Patients then receive 6 cycles of post-Consolidation therapy starting at least 1 week following radiation therapy, including sargramostim, dinutuximab, and isotretinoin.
Period: Overall Study
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Started | 42
Completed | 22
Not Completed | 20
Not completed — Death | 1
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 7
Not completed — Patient/Parent Refusal | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 3.4 [0.3 to 17.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 22
  More than one race | 1
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 30
  Australia | 7
  New Zealand | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Unacceptable Toxicity
Description: Assessed with National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Assessed by estimation of the combined toxic death and unacceptable toxicity rate during Induction cycles 3-5 together with a 95% confidence interval.
Time Frame: Up to the first 5 cycles of treatment
Population: All eligible patients who received at least one dose of ch14.18 (dinutuximab) during Induction cycles
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Number analyzed (Participants) | 42
percentage of patients | 0.0 [0.0 to 0.0]

2. Primary Outcome: Percentage of Participants Who Are Feasibility "Failure"
Description: Feasibility "failures" were defined as patients that did not receive >= 75% of the planned dinutuximab doses during Induction cycles 3-5. Assessed by estimation of the feasibility "failure" rate together with a 95% confidence interval.
Time Frame: Up to the first 5 cycles of treatment
Population: All eligible patients who received at least one dose of ch14.18 (dinutuximab) during Induction cycles
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Number analyzed (Participants) | 42
Percentage of patients | 0.0 [0.0 to 0.0]

3. Secondary Outcome: Response Rate
Description: Per the revised INRC, response is comprised by responses in 3 components: primary tumor, soft tissue and bone metastases, and bone marrow. Primary and metastatic soft tissue sites were assessed using Response Evaluation Criteria in Solid Tumors and MIBG scans or FDG-PET scans if the tumor was MIBG non-avid. Bone marrow was assessed by histology or immunohistochemistry and cytology or immunocytology. Complete response (CR) - All components meet criteria for CR. Partial response (PR) - PR in at least one component and all other components are either CR, minimal disease (in bone marrow), PR (soft tissue or bone) or not involved (NI; no component with progressive disease (PD). Minor response (MR) - PR or CR in at least one component but at least one other component with stable disease; no component with PD. Stable disease (SD) - Stable disease in one component with no better than SD or NI in any other component; no component with PD. Progressive disease (PD) - Any component with PD.
Time Frame: Up to the first 5 cycles of treatment
Population: All eligible patients. Institutional assessment of end-induction response has been used.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Number analyzed (Participants) | 42
Percentage of patients | 78.6 [64.1 to 88.3]

4. Secondary Outcome: Event-free Survival
Description: Per the revised INRC, progressive disease is: 1) > 20% increase in the longest diameter of the primary tumor, taking as reference the smallest sum and ¬> increase of 5 mm in longest dimension, 2) Any new soft tissue lesion detected by CT/MRI that is MIBG avid or FDG-PET avid, 3) Any new soft tissue lesion seen on CT/MRI that is biopsied and found to be neuroblastoma or ganglioneuroblastoma, 4) Any new bone site that is MIBG avid, 5) Any new bone site that is FDG-PET avid and has CT/MRI findings of tumor or is histologically neuroblastoma or ganglioneuroblastoma 6) A metastatic soft tissue site with > 20% increase in longest diameter, taking as reference the smallest sum on study, and with > 5mm in sum of diameters of target soft tissue lesions, 7) A relative MIBG score ¬> 1.2, 8) Bone marrow without tumor infiltration that becomes >5% tumor infiltration, 9) Bone marrow with tumor infiltration that increases by > 2-fold and has > 20% tumor infiltration on reassessment.
Time Frame: Up to 1 year
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Number analyzed (Participants) | 42
Percent Probability | 82.6 [70.8 to 94.4]

5. Secondary Outcome: Overall Survival
Description: Kaplan-Meier method was used to estimate overall survival (OS). OS was defined as the time from study enrollment to death. 1-year OS is provided.
Time Frame: Up to 1 year
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
Number analyzed (Participants) | 42
Percent Probability | 95.0 [88.1 to 100.0]

6. Other Pre Specified Outcome: Incidence of Naturally Occurring Anti-glycan Antibodies
Description: The Incidence of Naturally Occurring Anti-glycan Antibodies was calculated, including placement of a 95% CI on the incidence. In addition, anti-glycan levels prior to the start of Induction therapy and prior to the start of post-Consolidation therapy was compared with Wilcoxon's signed-rank test for paired data.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Incidence of Natural Killer (NK) Receptor NKp30 Isoforms
Description: Assessed by calculating the incidence of NK receptor NKp30 isoforms, including placement of a 95% CI on the incidence.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Response of Host Factors, Including Naturally Occurring Anti-glycan Antibodies, KIR/KIR-L Genotyping, Fc Receptor Genotyping, Human Anti-chimeric Antibodies (HACA)
Description: Explored with Fisher's exact test for categorical and Wilcoxon rank-sum test for continuous host factors. Both the presence/absence and level of naturally occurring anti-glycan antibodies was considered. For the KIR/KIR-L analysis, patients were categorized as either matched or mismatched. Patients were grouped into one of the three genotype subgroups of Fc receptor genotyping for that analysis. The presence/absence of HACA, anti-idiotype, and pretreatment anti-therapeutic antibodies (PATA)/anti-allotype antibody was considered for the HACA analysis.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Immune Environment (Gene Expression; Immune Effector Cells, Activities and Signaling Molecules; Immune Target Expression)
Description: The incidence of NK receptor NKp30 isoforms was calculated, including placement of a 95% CI on each incidence rate. Summary statistics were generated for serum cytokine (IL6, CXCL9) levels and gene expression of circulating immune function cells.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Levels of Circulating GD2 and Tumor Cell GD2 Expression
Description: Assessed by exploring the relationship between response to treatment with > PR (response vs. non- response) with circulating GD2 levels, and GD2 tumor cell expression following therapy with a Wilcoxon rank-sum test. Changes from baseline were also analyzed.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on Protocol Therapy, an average of 12 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT)
All-Cause Mortality (participants affected / at risk) | 1/42
Serious Adverse Events (participants affected / at risk) | 14/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT) (N=42)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Ascites (Gastrointestinal disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Chylous ascites (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
GGT increased (Investigations) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 2
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Ileus (Gastrointestinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Small intestinal mucositis (Gastrointestinal disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment(Chemotherapy, Dinutuximab, Sargramostim, ASCT, EBRT) (N=42)
Abdominal pain (Gastrointestinal disorders) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Anal mucositis (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 6
Anorectal infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 21
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 8
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Catheter related infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 3
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Dental caries (Gastrointestinal disorders) | 1
Device related infection (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 6
Enterocolitis infectious (Infections and infestations) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Eye infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 32
Fever (General disorders) | 21
Fungemia (Infections and infestations) | 2
GGT increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 15
Hematuria (Renal and urinary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Infections and infestations - Other, specify (Infections and infestations) | 9
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1
Jejunal obstruction (Gastrointestinal disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lethargy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 6
Malabsorption (Gastrointestinal disorders) | 1
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 31
Nausea (Gastrointestinal disorders) | 9
Neutrophil count decreased (Investigations) | 6
Pain (General disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2
Platelet count decreased (Investigations) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rectal mucositis (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 16
Shingles (Infections and infestations) | 2
Sinus tachycardia (Cardiac disorders) | 5
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 2
Small intestinal mucositis (Gastrointestinal disorders) | 2
Splenic infection (Infections and infestations) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Thrush (Infections and infestations) | 3
Thyroid stimulating hormone increased (Investigations) | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Typhlitis (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Viremia (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 11
Vulval infection (Infections and infestations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT03786783/Prot_SAP_000.pdf